CLINICAL TRIAL: NCT00045994
Title: Systolic and Pulse Pressure Hemodynamic Improvement By Restoring Elasticity: The SILVER Study
Brief Title: The SILVER Study: Systolic Hypertension Interaction With Left Ventricular Remodeling
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synvista Therapeutics, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALT-711-0107-Silver
Record Dates: First submitted 2002-09-17; First posted 2002-09-19 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2007-08

CONDITIONS: Hypertension; Hypertrophy, Left Ventricular
Keywords: cardiovascular; aged; antihypertensive agents/therapeutic use; hypertension/*drug therapy; blood pressure
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular | interventions — alagebrium

INTERVENTIONS:
Drug: ALT-711

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ALT-711 in the treatment of isolated systolic hypertension in a formal study in patients with left ventricular hypertrophy. Eligible patients will be randomized to double-blind treatment once daily for 6 months with oral ALT-711 (210 mg) or placebo.

ELIGIBILITY:
Inclusion Criteria

* Men or women at least 50 years of age.
* Screening diagnosis of isolated systolic hypertension, defined as systolic blood pressure >150 mm Hg and diastolic blood pressure <90 mm Hg (office blood pressure measurements) and systolic blood pressure >140 mm Hg (measured by 24-hour ambulatory blood pressure monitoring-mean daytime values).
* Baseline systolic blood pressure >150 mm Hg and diastolic blood pressure <90 mm Hg (office blood pressure measurements).
* Patients with left ventricular hypertrophy (LVH) as determined by limited echocardiography for LVH (i.e., wall thickness > 1.2 cm).
* Patient can complete an informed consent.

Exclusion Criteria

* Patient <50 years of age.
* Patients on antihypertensive therapy with changes in dose in the last 1 month prior to the entry into the study.
* Hb A1c > 9%.
* Serum creatinine > 1.7mg/dL.
* History of ketoacidosis or uncontrolled diabetes within the last 2 years.
* History of congestive heart failure.
* History of stroke, or any sequelae of a transient ischemic attack, reversible ischemic neurologic defect, or stroke, within the last 12 months.
* History of acute myocardial infarction within 6 months prior to entry into the study.
* Any significant ECG abnormalities, including second degree AV-block or complete AV-block. Any known significant arrhythmia including atrial flutter, ventricular tachycardia, WPW-syndrome. Any hemodynamically significant valvular heart disease.
* Any significant systemic illnesses or medical condition that could lead to difficulty complying with the protocol.
* Screening or Baseline liver function tests SGOT and/or SGPT > 2.0 times the upper limits of central laboratory normal range.
* Use of systemic and/or inhaled corticosteroids (excluding topical corticosteroids).
* Any additional condition(s), which in the investigator's opinion would prohibit the patient from completing the study, or not be in the best interest of the patient.
* Use of any investigational drugs within 30 days prior to screening.
* Previous exposure to ALT-711.
* Known seropositivity for HIV or hepatitis C, or presence of hepatitis B surface antigen.
* Pregnancy or active breast-feeding. Female patients of childbearing potential (not postmenopausal for at least 5 years or surgically sterilized) must agree not to become pregnant during the duration of the study. Specifically, they must agree to use an appropriate contraceptive regimen. Acceptable regimens include abstinence, systemic hormones, intrauterine devices and barrier methods, such as cervical caps, male or female condoms, or diaphragms with concomitant intravaginal spermicide. A barrier method must have been used without failure for at least 1 year immediately preceding entry into the study.
* Positive drug screen.
* Necessity to use tobacco or nicotine-containing products, or to consume caffeine- containing beverages and/or food, and/or alcohol after midnight prior to clinic visit days, until after any evaluations.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2001-08; Primary Completion 2002-01 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milan Kovacevic, MD, PhD, Study Director — Synvista Therapeutics, Inc

REFERENCES:
- [Background] Kass DA, Shapiro EP, Kawaguchi M, Capriotti AR, Scuteri A, deGroof RC, Lakatta EG. Improved arterial compliance by a novel advanced glycation end-product crosslink breaker. Circulation. 2001 Sep 25;104(13):1464-70. doi: 10.1161/hc3801.097806. PMID 11571237
- [Background] Asif M, Egan J, Vasan S, Jyothirmayi GN, Masurekar MR, Lopez S, Williams C, Torres RL, Wagle D, Ulrich P, Cerami A, Brines M, Regan TJ. An advanced glycation endproduct cross-link breaker can reverse age-related increases in myocardial stiffness. Proc Natl Acad Sci U S A. 2000 Mar 14;97(6):2809-13. doi: 10.1073/pnas.040558497. PMID 10706607
- [Background] Wolffenbuttel BH, Boulanger CM, Crijns FR, Huijberts MS, Poitevin P, Swennen GN, Vasan S, Egan JJ, Ulrich P, Cerami A, Levy BI. Breakers of advanced glycation end products restore large artery properties in experimental diabetes. Proc Natl Acad Sci U S A. 1998 Apr 14;95(8):4630-4. doi: 10.1073/pnas.95.8.4630. PMID 9539789
- [Background] Vaitkevicius PV, Lane M, Spurgeon H, Ingram DK, Roth GS, Egan JJ, Vasan S, Wagle DR, Ulrich P, Brines M, Wuerth JP, Cerami A, Lakatta EG. A cross-link breaker has sustained effects on arterial and ventricular properties in older rhesus monkeys. Proc Natl Acad Sci U S A. 2001 Jan 30;98(3):1171-5. doi: 10.1073/pnas.98.3.1171. PMID 11158613
- [Background] Chobanian AV. Control of hypertension--an important national priority. N Engl J Med. 2001 Aug 16;345(7):534-5. doi: 10.1056/NEJM200108163450709. No abstract available. PMID 11519509
- [Background] Hyman DJ, Pavlik VN. Characteristics of patients with uncontrolled hypertension in the United States. N Engl J Med. 2001 Aug 16;345(7):479-86. doi: 10.1056/NEJMoa010273. PMID 11519501
- [Background] Wilkinson IB, Webb Christison DJ, Cockcroft JR. Isolated systolic hypertension: a radical rethink. It's a risk factor that needs treatment, especially in the over 50s. BMJ. 2000 Jun 24;320(7251):1685. doi: 10.1136/bmj.320.7251.1685. No abstract available. PMID 10864525
- [Background] Brownlee M, Vlassara H, Kooney A, Ulrich P, Cerami A. Aminoguanidine prevents diabetes-induced arterial wall protein cross-linking. Science. 1986 Jun 27;232(4758):1629-32. doi: 10.1126/science.3487117.
- [Background] McVeigh GE, Bratteli CW, Morgan DJ, Alinder CM, Glasser SP, Finkelstein SM, Cohn JN. Age-related abnormalities in arterial compliance identified by pressure pulse contour analysis: aging and arterial compliance. Hypertension. 1999 Jun;33(6):1392-8. doi: 10.1161/01.hyp.33.6.1392. PMID 10373222
- [Background] Neaton JD, Wentworth D. Serum cholesterol, blood pressure, cigarette smoking, and death from coronary heart disease. Overall findings and differences by age for 316,099 white men. Multiple Risk Factor Intervention Trial Research Group. Arch Intern Med. 1992 Jan;152(1):56-64. PMID 1728930